CLINICAL TRIAL: NCT04681222
Title: Postoperative Pain Management in Patients Undergoing Total Hip Arthroplasty: PENG Block in Combination With LFCN Block or Wound Infiltration?
Brief Title: Comparison of the Efficacy of PENG Block in Combination With LFCN Block and Wound Infiltration
Status: Completed | Type: Observational
Sponsor: Derince Training and Research Hospital (Other)
Collaborators: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Hande Gurbuz, Medical Doctor, Associate Professor, Principal Investigator, Derince Training and Research Hospital
Other Study IDs: U1111-1262-9877
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Postoperative Pain
Keywords: Coxarthrosis; Regional Anesthesia; Total Hip Replacement
MeSH Terms: conditions — Pain, Postoperative; Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LFCN: Patients received LFCN + PENG blocks
  Interventions: Procedure: LFCN
- Wound Infiltration: Patients received wound infiltration + PENG blocks
  Interventions: Procedure: Wound infiltration

INTERVENTIONS:
Procedure: LFCN — LFCN block was performed in combination with PENG block
  Groups: LFCN
Procedure: Wound infiltration — Wound infiltration was performed in combination with PENG block
  Groups: Wound Infiltration

SUMMARY:
The ultrasound-guided approach for the blockade of articular branches of femoral and obturator nerves, pericapsular nerve group (PENG) block, is an effective method for postoperative analgesia in hip surgeries.

DETAILED DESCRIPTION:
The ultrasound-guided approach for the blockade of articular branches of femoral and obturator nerves, pericapsular nerve group (PENG) block, is an effective method for postoperative analgesia in hip surgeries. However, it fails to provide cutaneous analgesia on the anterolateral surgical incisional site. This study compares the effects of wound infiltration and lateral femoral nerve blocks in combination with PENG blocks for postoperative pain in patients undergoing total hip arthroplasty for coxarthrosis.

ELIGIBILITY:
Inclusion Criteria:

* Coxarthrosis
* Total hip replacement
* Patients agreed to receive PENG block
* LFCN or wound infiltration performed combined with PENG blocks

Exclusion Criteria:

* Other kinds of hip surgeries
* Total hip replacement performed for other indications
* Patients refused to receive PENG block

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients underwent total hip arthroplasty with the diagnosis of coxarthrosis, and those received PENG blocks for postoperative analgesia combined with whether LFCN block or wound infiltration.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
First analgesic demand | 24 hours
  The time interval from PENG blocks to the first analgesic demand.

SECONDARY OUTCOMES:
Opioid consumption | 24 hours
  Total opioid analgesic consumption
Numeric Rating Scale | 24 hours
  The maximum score on a 10cm numeric rating scale: (0 to 10cm) (0 = no pain, 10 = worst imaginable pain)
Nonsteroidal Anti-inflammatory Drugs (NSAID) | 24 hours
  Total NSAID consumption

CONTACTS AND LOCATIONS:
Locations (1):
- Derince Training and Research Hospital, Kocaeli, Derince, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Background] Roy R, Agarwal G, Pradhan C, Kuanar D. Total postoperative analgesia for hip surgeries, PENG block with LFCN block. Reg Anesth Pain Med. 2019 Mar 28:rapm-2019-100454. doi: 10.1136/rapm-2019-100454. Online ahead of print. No abstract available. PMID 30923252
- [Background] Nersesjan M, Hagi-Pedersen D, Andersen JH, Mathiesen O, Dahl JB, Broeng L, Thybo KH. Sensory distribution of the lateral femoral cutaneous nerve block - a randomised, blinded trial. Acta Anaesthesiol Scand. 2018 Jul;62(6):863-873. doi: 10.1111/aas.13091. Epub 2018 Feb 21. PMID 29468642
- [Background] Giron-Arango L, Roques V, Peng P. Reply To Dr Roy et al: Total postoperative analgesia for hip surgeries: PENG block with LFCN block. Reg Anesth Pain Med. 2019 Mar 28:rapm-2019-100505. doi: 10.1136/rapm-2019-100505. Online ahead of print. No abstract available. PMID 30923249
- [Background] Mistry T, Sonawane KB, Kuppusamy E. PENG block: points to ponder. Reg Anesth Pain Med. 2019 Mar;44(3):423-424. doi: 10.1136/rapm-2018-100327. Epub 2019 Jan 11. No abstract available. PMID 30635514